CLINICAL TRIAL: NCT03430531
Title: Effectiveness of Sphenopalatine Ganglion Block for Post-Dural Puncture Headache; A Pilot Study
Brief Title: Effectiveness of Sphenopalatine Ganglion Block for Post-Dural Puncture Headache
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study suspended and subsequently terminated due to Pandemic
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Verghese T Cherian, MD, Associate Professor of Anesthesiology & Perioperative Medicine, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8426
Record Dates: First submitted 2018-02-06; First posted 2018-02-13 (Actual); Results first posted 2022-06-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-05

CONDITIONS: Post-Dural Puncture Headache; Sphenopalatine Ganglion Block
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: Open-label, single arm, pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sphenopalatine ganglion block (Experimental): Sphenopalatine ganglion block: this block will be performed by inserting swabs, with lidocaine squirted on them, into each nostril and reaching the nasopharyngeal wall.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Lidocaine 2% viscous (0.5ml) will be squirted on two cotton swab sticks and one will be gently inserted into each nostril, along the floor of the nose. Slight rotatory motion of the stick will be used to insert it as far as it goes with the intention to reach the nasopharyngeal wall (posterior wall of the nose). At that position the swab sticks will be left undisturbed for 5 minutes. The swabs will be taken out and this will be repeated twice more, using fresh swabs and 0.5ml of 2% lidocaine. The block would take about 30 minutes.

SUMMARY:
The objective of the study is to determine the effectiveness of Spheno-Palatine (SP) ganglion block to alleviate the pain of post-dural puncture headache (PDPH).

DETAILED DESCRIPTION:
The primary objectives of the study are to study the effectiveness of SP ganglion block in relieving post-dural puncture headache in terms of :

1. Number of subjects who get relief of pain
2. The onset time to pain relief after application of block
3. The duration of pain relief
4. The incidence of recurrence of post-dural puncture headache

Secondary objectives are to:

1. Monitor any complications due to SP ganglion block
2. Measure patient satisfaction
3. Monitor any residual effects at 1 months after the SP block

ELIGIBILITY:
Inclusion Criteria:

1. Complains of symptoms suggestive of post-dural puncture headache
2. Has a history of dural puncture (lumbar puncture or accidental dural puncture during epidural placement) within the previous 7 days
3. Fluent in written and spoken English

Exclusion Criteria:

1. Those with a known history of hypersensitivity to local anesthetics of the amide type or to other components of GLYDO
2. Those with any congenital or acquired, anatomical deformity of the nostril, which preclude performing the block
3. Those who refuse to consent to participate in the study
4. Patients who have had a failed epidural blood patch
5. Cognitive Impairment
6. Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2022-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Verghese Cherian, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sphenopalatine Ganglion Block
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sphenopalatine Ganglion Block
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Pain Score at Baseline
Description: Pain scores will be recorded at Baseline in a sitting position. Pain scores will be quantified using the Visual analog pain (VAS) scale. The visual analog scale (VAS) is a tool widely used to measure pain. The scale range is 0-10 with 0 being no pain and 10 being severe pain.
Time Frame: 15 minutes before the SP block
Population: Subjects receiving a Sphenopalatine ganglion block for treatment of a severe post-epidural spinal headache.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sphenopalatine Ganglion Block
Number analyzed (Participants) | 6
units on a scale | 9.33 (0.82)

2. Primary Outcome: Pain Score 60 Minutes Post-SP Block
Description: Pain scores will be recorded 60 minutes post-SP block in a sitting position. Pain scores will be quantified using the Visual analog pain (VAS) scale. The visual analog scale (VAS) is a tool widely used to measure pain. The scale range is 0-10 with 0 being no pain and 10 being severe pain.
Time Frame: 60 minutes
Population: Subjects receiving a Sphenopalatine ganglion block for treatment of a severe post-epidural spinal headache.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sphenopalatine Ganglion Block
Number analyzed (Participants) | 6
units on a scale | 0.33 (0.82)

3. Primary Outcome: Pain Score 1 Day Post-SP Block
Description: Patient reported pain scores will be recorded day 1 post SP block in a sitting position. Pain scores will be quantified using the Visual analog pain (VAS) scale. The visual analog scale (VAS) is a tool widely used to measure pain. The scale range is 0-10 with 0 being no pain and 10 being severe pain.
Time Frame: 1 day
Population: Subjects receiving a Sphenopalatine ganglion block for treatment of a severe post-epidural spinal headache.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sphenopalatine Ganglion Block
Number analyzed (Participants) | 6
units on a scale | 5.33 (3.50)

4. Primary Outcome: Pain Score 2 Days Post-SP Block
Description: Patient reported pain scores will be recorded day 2 post SP block in a sitting position. Pain scores will be quantified using the Visual analog pain (VAS) scale. The visual analog scale (VAS) is a tool widely used to measure pain. The scale range is 0-10 with 0 being no pain and 10 being severe pain.
Time Frame: 2 days
Population: Subjects receiving a Sphenopalatine ganglion block for treatment of a severe post-epidural spinal headache.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sphenopalatine Ganglion Block
Number analyzed (Participants) | 6
units on a scale | 3.67 (2.66)

5. Primary Outcome: Pain Score 7 Days Post-SP Block
Description: Patient reported pain scores will be recorded day 7 post SP block in a sitting position. Pain scores will be quantified using the Visual analog pain (VAS) scale. The visual analog scale (VAS) is a tool widely used to measure pain. The scale range is 0-10 with 0 being no pain and 10 being severe pain.
Time Frame: 7 days
Population: Subjects receiving a Sphenopalatine ganglion block for treatment of a severe post-epidural spinal headache.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sphenopalatine Ganglion Block
Number analyzed (Participants) | 6
units on a scale | 2.33 (1.97)

6. Primary Outcome: Pain Score 30 Day Post-SP Block
Description: Patient reported pain scores will be recorded day 30 post SP block in a sitting position. Pain scores will be quantified using the Visual analog pain (VAS) scale. The visual analog scale (VAS) is a tool widely used to measure pain. The scale range is 0-10 with 0 being no pain and 10 being severe pain.
Time Frame: 30 days
Population: Subjects receiving a Sphenopalatine ganglion block for treatment of a severe post-epidural spinal headache.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sphenopalatine Ganglion Block
Number analyzed (Participants) | 6
units on a scale | 1.67 (1.37)

7. Secondary Outcome: Duration of Pain Relief
Description: Patient reported how long after the SP block the patient reported pain scores that were decreased form the baseline measures. The outcome measure is measured in hours that pain relief was achieved.
Time Frame: 24 hours
Population: Subjects who received an SP block for treatment of a severe post-epidural headache who did not see complete resolution of their pain.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Sphenopalatine Ganglion Block
Number analyzed (Participants) | 4
hours | 13.50 (4.43)

8. Secondary Outcome: Number of Participants With Recurrence of Post-dural Puncture Headache
Description: Patient reported recurrence of post dural puncture headache resulting in treatment with epidural blood patch
Time Frame: 7 days
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Sphenopalatine Ganglion Block
Number analyzed (Participants) | 6
Participants | 4

9. Secondary Outcome: Number of Participants With Complications Due to SP Ganglion Block
Description: Patients will be asked to report any side effects, including: allergic reaction to lidocaine, nose irritation and nose-bleed.
Time Frame: 15 minutes before the SP block to 30 days post SP block
Population: Subjects receiving a Sphenopalatine ganglion block for treatment of a severe post-epidural spinal headache.
Measure: Count of Participants; unit: Participants
Arm/Group | Sphenopalatine Ganglion Block
Number analyzed (Participants) | 6
Participants | 0

ADVERSE EVENTS:
Time Frame: Subjects were monitored for any adverse events for 30 days post-SP block.
Arm/Group | Sphenopalatine Ganglion Block
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
The target enrollment was not reached secondary to the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/31/NCT03430531/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/31/NCT03430531/ICF_001.pdf